CLINICAL TRIAL: NCT07090681
Title: Novel Individualized Brain Stimulation, Network-based Approaches to Improve Cognition in Healthy Seniors and Patients With MCI
Brief Title: Novel Individualized Brain Stimulation, Network-based Approaches to Improve Cognition in Healthy Seniors and MCI Patients
Acronym: NIBS-iCOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (EPFL), Campus Biotech (Unknown); Masaryk University (Other)
Responsible Party: Principal Investigator, Friedhelm Hummel, Professor, Ecole Polytechnique Fédérale de Lausanne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-00127-wp10; 320030L_197899 (Other Grant/Funding Number: SNSF)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment (MCI); Healthy Aging
Keywords: NIBS; tTIS; MCI; aMCI; LB-MCI; TMS; iTBS; striatum; cerebellum
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild Cognitive Impairment (Experimental): Patients with mild cognitive impairment
  Interventions: Device: Active Control Placebo; Device: tTIS; Device: tTIS + TMS
- Healthy Elderly (Active Comparator): Cognitively Unimpaired individuals older than 60 years
  Interventions: Device: Active Control Placebo; Device: tTIS; Device: tTIS + TMS

INTERVENTIONS:
Device: Active Control Placebo — In this intervention, participants underwent magnetic stimulation at the neck level with a TMS coil. Ten minutes after, they received a high frequency temporal interference stimulation with an overlapping sinusoidal wave at 2KHz, without any interferent pattern.
Device: tTIS — In this intervention, participants underwent magnetic stimulation at the neck level with a TMS coil. Ten minutes after, they received active transcranial temporal interference stimulation with a patterned stimulation (intermittent theta-burst) generating temporal interference in the striatum; see Wessel et al., 2023, Nat Neurosci. for details
Device: tTIS + TMS — In this intervention, participants underwent cerebellar magnetic stimulation at the level of a predefined individual point in the inferior left cerebellar hemisphere with a TMS coil, receiving a total of 600 pulses organised in an intermittent theta-burst pattern. Ten minutes after, they received active transcranial temporal interference stimulation with a patterned stimulation (intermittent theta-burst) generating temporal interference in the striatum; see Wessel et al., 2023, Nat Neurosci. for details

SUMMARY:
Working memory (WM) relies on a vast network comprising cortical and subcortical structures and its impairment is frequent in normal aging, mild cognitive impairment (MCI) and dementia, often driving fucntional decline. Recent studies have shown that non-invasive brain stimulation (NIBS) methods can modulate neuronal activity, and brain network interactions. A significant body of literature has shown that both striatum and cerebellum are reciprocally connected and implicated in WM performance. However, to date, NIBS studies have mainly focused on cerebellar stimulation with transcranial magnetic stimulation (TMS), often yielding inconclusive or conflicting results. In the investigator hypothesis, sequential and concurrent stimulation of multiple brain regions of the WM subcortical network (i.e. targeting striatum and cerebellum) via transcranial temporal interference stimulation (tTIS) and/or repetitive transcranial magnetic stimulation (rTMS) could enhance WM performance in healthy elderly and/or MCI patients. Moreover, combining different stimulation techniques with multimodal neuroimaging and computational modeling, the investigators expect to acquire better mechanistic understanding through which different NIBS act on the brain and improves cognitive functions.

DETAILED DESCRIPTION:
Executive functions and particularly working memory (WM) play a crucial role in daily life and is frequently impaired in patients with mild cognitive impairment (MCI), constituting one of the driving factors that compromise quality of life and autonomy. WM specifically relies on a vast brain network of cortical and subcortical regions. Among the different subcortical structures implicated in executive functions, both striatum and cerebellum have been linked to WM performance with complementary roles. Striatum is variably affected in the course of different neurodegenerative diseases, while in contrast, the cerebellum has been associated with cognitive resilience and brain reserve, making it a promising target for interventions for cognitive enhancement.

Hence, leveraging the reciprocal striato-cerebellar connections, in this multi-center, randomized, placebo-controlled proof-of-concept trial, the investigators implemented a sequential multifocal plasticity-inducing stimulation of the striatum and the cerebellum to enhance WM in MCI patients.

The investigators will apply an excitatory intermittent theta burst (iTBS) cerebellar TMS to target the left inferior cerebellar hemisphere and transcranial temporal interference stimulation (tTIS) with the same pattern to focally neuromodulate the striatum in MCI patients. In our hypothesis, this combined sequential protocol will synergistically enhance WM performance.

The investigators will analyse not only the resulting behavioral data as the main outcome, but via multimodal neuroimaging (structural and functional magnetic resonance imaging; s/fMRI) and computational modeling methods they will dissect the network mechanisms and patterns of intrinsic connectivity changes underlying the behavioral changes.

ELIGIBILITY:
Inclusion Criteria:

* For MCI:
* Age > 18 years old;
* Clinical diagnosis of MCI due to possible or probable Lewy Bodies Dementia or amnestic MCI following core clinical and neuropsychological criteria.
* For Healthy Elderlies:
* Age > 60 years old;
* Normal performance on baseline cognitive screening.

Exclusion Criteria:

* presence of dementia as assessed by a cognitive test battery and evaluation of daily activities, any major psychiatric disorder (including major depressive episode);
* history of another neurological disease affecting central nervous system (e.g., tumor, epilepsy, stroke, etc.);
* severe or repeated head injury;
* non-compensated systemic or oncological disease;
* presence of MRI-incompatible metal in the body (e.g., cardiac pacemaker).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Working memory performance | through study completion, an average of 1 year
  The investigators will compare the baseline-normalized reaction time (in milliseconds) and error rate (number of correct and incorrect responses) of a visual working memory task between the active tTIS and tTIS and TMS and the placebo stimulation condition in a cross-over design.

SECONDARY OUTCOMES:
The neural underpinnings of NIBS-induced changes quantified by s/fMRI and network-based analytical approaches. | The changes will be computed from the difference between connectivity at baseline and 1 hour post-stimulation.
  The changes in intra- and inter-regional fMRI connectivity (measured by BOLD signal variations in specific brain regions expressed as z-scores) within and between cognitive brain networks will be compared between the active inerventions (tTIS and tTIS+TMS) and the active control stimulations.

CONTACTS AND LOCATIONS:
Overall Officials: Friedhelm Cristoph Hummel, Professor, Principal Investigator — Defitech Chair of Clinical Neuroengineering, Neuro-X Institute (INX), École Polytechnique Fédérale de Lausanne (EPFL); Irena Rektorova, Professor, Principal Investigator — Neuroscience Program, Central European Institute of Technology, Masaryk University, Brno, Czech Republic
Locations (2):
- CEITEC, Brno, Czechia
- Campus Biotech, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided